CLINICAL TRIAL: NCT01702233
Title: Treatment of Rotator Cuff Syndrome and Bursitis: A Double Blind, Controlled Trial to Assess the Efficacy and Safety of Traumeel® S Injection Versus Corticosteroid Injections and Versus Placebo
Brief Title: TRARO (Traumeel® S in Rotator Cuff Syndrome)-Study
Acronym: TRARO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biologische Heilmittel Heel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRARO; 2012-003393-12 (EudraCT Number)
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Rotator Cuff Syndrome; Shoulder Bursitis
MeSH Terms: interventions — Traumeel S; dexamethasone acetate; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Traumeel S inj. (Experimental): Traumeel S inj. 2 ml. subacromial 3 times at days 1, 8 and 15
  Interventions: Drug: Traumeel S inj
- Fortecortin/Dexamethasone 8 mg inj (Active Comparator): Fortecortin/Dexamethasone 8 mg/2 ml inj. subacromial 3 times at days 1, 8 and 15
  Interventions: Drug: Fortecortin/Dexamethasone 8 mg/2 ml inj
- Saline inj. (Placebo Comparator): Saline inj. 2 ml. subacromial 3 times at days 1, 8 and 15
  Interventions: Drug: Saline inj

INTERVENTIONS:
Drug: Traumeel S inj — Traumeel S inj. 2 ml. subacromial 3 times at days 1, 8 and 15
  Other Names: Traumeel
  Arms: Traumeel S inj.
Drug: Fortecortin/Dexamethasone 8 mg/2 ml inj — Fortecortin/Dexamethasone 8 mg/2 ml inj. subacromial 3 times at days 1, 8 and 15
  Other Names: Dexamethasone 8 mg
  Arms: Fortecortin/Dexamethasone 8 mg inj
Drug: Saline inj — Saline inj. 2 ml. subacromial 3 times at days 1, 8 and 15
  Other Names: Placebo inj
  Arms: Saline inj.

SUMMARY:
To evaluate functional, clinical, and subjective parameters in patients with rotator cuff syndrome and bursitis treated with Traumeel® S injections versus corticosteroid injections and versus placebo. 160 patients are planned to be randomised (i.e., 64 patients per active treatment group and 32 patients in the placebo group) in 9 investigator sites in Germany, Belgium and Spain.

Finally 176 patients have been randomized (73 Traumeel, 67 Fortecortin and 36 Placebo) and 175 of them received at least one dosage of treatment

DETAILED DESCRIPTION:
Duration of the study were 16 weeks. Duration of Treatments were 15 days, applying one injection of 2 ml od study medication at days 1, 8, and 15. There was a follow up visit at day 22 (Primary endpoint), a telephone visit at week 9 and a final visit at week 15.

Standard descriptive summary statistics were calculated for continuous variables (i.e. arithmetic mean, standard deviation, minimum value, median, maximum value, number of non-missing values). All statistical analyses in this study were of exploratory nature. The summaries of the efficacy parameters, the statistical analyses of the primary efficacy variable, and the statistical analyses of the secondary efficacy variables were performed on the PP Set. These summaries and analyses were supported by corresponding summaries and exploratory statistical analyses performed on the Full Analysis Set. Missing values for all efficacy parameters were imputed by the last observation carried forward (LOCF) approach. The Modified Per-Protocol (MPP) Set excluded from the PP Set also all patients having taken unallowed concomitant medication after Visit 5 and was used as a secondary population for the analysis of efficacy. All statistical tests were two-sided with a significance level of (alpha) = 0.05, unless specified otherwise. The primary efficacy variable was the change from baseline in VAS for abduction rotation pain at Visit 5 (Day 22) (Traumeel® S injections versus corticoid injections) for active external rotation.

A one-sided test of non-inferiority of Traumeel® S with respect to dexamethasone at level 0.025 was computed using an analysis of covariance (ANCOVA) model with treatment group as qualitative factor and the baseline value of the abduction rotation pain VAS for active external rotation as a covariate. The test decision was based on a one-sided 97.5% confidence interval for the corresponding treatment difference. The non-inferiority margin was set to 13 mm on a 0 - 100 mm VAS scale.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with acute episodes of chronic rotator cuff syndrome and/or bursitis: tendinopathy of the supraspinatus tendon, bursitis, or partial degenerative tears of the supraspinatus and/or infraspinatus tendon (differentiation by ultrasonography)
2. Age 40 to 65 years, inclusive
3. Willing and able to understand and sign an approved informed consent form
4. Not pregnant (as proven by negative pregnancy test before first study drug administration) or breast-feeding. Females of childbearing potential (including those less than one year post-menopausal) must agree to maintain reliable birth control throughout the study, i.e. an established use of oral, injected or implanted hormonal contraception, female sterilization by hysterectomy, bilateral oophorectomy, or bilateral tubal exeresis, intrauterine device ([IUD] or coil or barrier method (e.g. diaphragm, cervical/vault cap) plus spermicidal cream/gel

Exclusion Criteria:

1. Calcifications in shoulder joint
2. Complete rotator cuff tears
3. Treatment with non-steroidal anti-inflammatory drugs (NSAIDs). Previous treatment with NSAIDs is allowed, with a wash-out period of 1 week; paracetamol can be taken until 48 hours before baseline visit
4. Corticoid therapy by mouth or by injection within the previous 3 months prior to screening
5. Any contraindication for corticoid therapy
6. Physical Therapy, acupuncture, transcutaneous electrical nerve stimulation (TENS) and shock-wave therapy (within 30 days prior to screening)
7. Treatment with anticoagulants (except low-dose aspirin)
8. Diabetic patients including borderline cases (glycosylated fraction of hemoglobin [HbA1c] > 7.0% at screening)
9. Clinically significant shoulder joint deformities
10. Major injury, including sports-related injury, to the shoulder within the past year
11. Significant osteoarthritis of the shoulder
12. Cervical spine disorder (that could confound the clinical assessment) that has been symptomatic and required active treatment within the past three months before screening
13. Any active musculoskeletal disease that could confound the diagnosis/evaluation of the painful shoulder, any neurological aetiology of the pain, or any acute infection of the shoulder joint
14. Any major surgery, arthroplasty, or arthroscopy in the signal shoulder within 6 months of screening or planned surgery within the duration of the study
15. Prior history of any malignancy (with the exception of basal cell carcinoma) treated less than 2 years ago
16. Patients with rheumatic polymyalgia
17. Known or suspected allergies against one or any particular ingredients of Traumeel® S or of other study preparations
18. Presence of serious gastrointestinal, renal, hepatic, pulmonary, cardiovascular, neurological disease or other known systemic disease (like leukemia, tuberculosis, immune mediated diseases, multiple sclerosis, Acquired Immuno Deficiency Syndrome, Human Immunodeficiency Virus-infections or other chronic virus-infections) that might interfere with the outcome of the study or the patient's ability to comply with study requirements.
19. Presence of infections and/or skin diseases in the area of the injection site (including psoriasis)
20. Clinically significant abnormal laboratory values (as judged of the investigator) at the screening visit
21. Consumption of any investigational product within one month prior to the screening visit
22. Patients who are likely to be non-compliant or uncooperative during the study, as judged by the investigator.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luc Vandenbossche, MD, PhD, Principal Investigator — Physical and Rehabilitation Medicine University Ghent, BE
Locations (1):
- Luc Vandenbossche, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vanden Bossche L, Vanderstraeten G. A multi-center, double-blind, randomized, placebo-controlled trial protocol to assess Traumeel injection vs dexamethasone injection in rotator cuff syndrome: the TRAumeel in ROtator cuff syndrome (TRARO) study protocol. BMC Musculoskelet Disord. 2015 Feb 4;16(1):8. doi: 10.1186/s12891-015-0471-z. PMID 25649543

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 176 patients have been randomized, 175 of them started treatment. 1 Patient in Treatment arm Traumeel S withdrew consent before first dose.
Period: Overall Study
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj | Saline Inj.
Started | 72 | 67 | 36
Full Analysis Set (ITT) | 66 | 63 | 31
Per Protocol Set | 58 | 58 | 27
Completed | 66 | 64 (One of these Patient completed the Trial but had no valid outcome measure after enrolment) | 31
Not Completed | 6 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj | Saline Inj. | Total
Number analyzed (Participants) | 72 | 67 | 36 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 72 | 67 | 36 | 175
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.00 (6.90) | 51.90 (7.02) | 51.80 (6.74) | 51.50 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 16 | 77
  Male | 41 | 37 | 20 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 72 | 66 | 35 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 5 | 2 | 2 | 9
  Germany | 52 | 51 | 25 | 128
  Spain | 15 | 14 | 9 | 38
Screening Height [Mean (Standard Deviation); unit: cm] | 171.3 (10.24) | 170.6 (8.01) | 169.9 (11.32) | 170.8 (9.65)
Screening Weight [Mean (Standard Deviation); unit: kg] | 76.4 (16.57) | 79.2 (14.90) | 78.8 (16.90) | 78 (15.98)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.92 (4.455) | 27.29 (5.455) | 27.14 (4.382) | 26.69 (4.866)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Abduction Rotation Pain VAS at Visit 5 (Day 22) (Traumeel® S Injections Versus Fortecortin) for Active External Rotation
Description: VAS is a 100 mm visual analogue scale for measuring the pain resulted from the adbuction and external rotation of the arm. Possible scores range from 0 (no pain) to 100 (worst possible pain). Change = (Day 22 score -- baseline score).
Time Frame: Baseline to Day 22
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale (mm)
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj
Number analyzed (Participants) | 58 | 58
units on a scale (mm) | -18.7 (21.49) | -27.2 (23.44)
Statistical Analysis 1: Comparison: Traumeel S Inj. vs Fortecortin/Dexamethasone 8 mg Inj; Test type: Non-Inferiority or Equivalence — All statistical analyses were of exploratory nature. A one-sided test of non-inferiority of Traumeel®S with respect to dexamethasone at level 0.025 was computed using an analysis of covariance (ANCOVA) model with treatment group as qualitative factor and the baseline value of the abduction rotation pain VAS for active external rotation as a covariate. The test decision was based on a one-sided 97.5% confidence interval . The non-inferiority margin was set to 13 mm on a 0-100 mm VAS scale; p < 0.05, ANCOVA; Mean Difference (Final Values) = 13, 95% CI 1-sided [upper limit 97.5], Standard Deviation 13

2. Secondary Outcome: Change From Baseline in Abduction Rotation Pain VAS for Active External Rotation - Comparison With Placebo Visit 5 (Day 22)
Description: VAS is a 100 mm visual analogue scale for measuring the pain resulted from the adbuction and external rotation of the arm. Possible scores range from 0 (no pain) to 100 (worst possible pain).
Time Frame: Baseline vs. Day 22
Measure: Mean (Standard Deviation); unit: Change in mm baseline vs. day 22
Arm/Group | Traumeel S Inj. | Saline Inj
Number analyzed (Participants) | 58 | 27
Change in mm baseline vs. day 22 | -18.7 (21.49) | -17.1 (23.94)

3. Secondary Outcome: Change From Baseline in Abduction Rotation Pain VAS for Active External Rotation - Comparison With Placebo Visit 7 (Day 105)
Description: as for outcome 2
Time Frame: Baseline vs. Day 105
Measure: Mean (Standard Deviation); unit: units on a scale, mm
Arm/Group | Traumeel S Inj. | Saline Inj
Number analyzed (Participants) | 58 | 27
units on a scale, mm | -32.2 (26.59) | -30.1 (27.80)

4. Secondary Outcome: Change From Baseline in Abduction Rotation Pain VAS for Active External Rotation - Comparison With Fortecortin at Visit 7 (Day 105)
Description: as for outcome 2
Time Frame: Baseline vs. day 105
Measure: Mean (Standard Deviation); unit: units on a scale, mm
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj
Number analyzed (Participants) | 58 | 58
units on a scale, mm | -32.2 (26.59) | -33.3 (28.35)

5. Secondary Outcome: Changes From Baseline in ROM in Degrees (Active External Rotation in Abduction) After Visit 5 (Day 22), Traumeel vs Placebo
Description: Range of movement (ROM) changes measured by active external rotation in abduction in degrees by goniometry in the range of 0 to 360 degrees.
Time Frame: Baseline vs. Day 22
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Traumeel S Inj. | Saline Inj
Number analyzed (Participants) | 58 | 27
degrees | 11.3 (15.73) | 13.5 (18.65)

6. Secondary Outcome: Changes From Baseline in ROM in Degrees (Active External Rotation in Abduction) After Visit 7 (Day 105), Traumeel vs Placebo
Description: as for outcome 5
Time Frame: Baseline vs. day 105
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Traumeel S Inj. | Saline Inj
Number analyzed (Participants) | 58 | 27
degrees | 13.9 (19.97) | 20.0 (20.19)

7. Secondary Outcome: Changes From Baseline in ROM in Degrees (Active External Rotation in Abduction) After Visit 5 (Day 22) Traumeel vs Fortecortin
Description: as for outcome 5
Time Frame: Baseline vs. Day 22
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj
Number analyzed (Participants) | 58 | 58
degrees | 11.3 (15.73) | 17.2 (21.03)

8. Secondary Outcome: Changes From Baseline in ROM in Degrees (Active External Rotation in Abduction) After Visit 7 (Day 105), Traumeel vs Fortecortin
Description: as for outcome 5
Time Frame: Baseline vs. Day 105
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj
Number analyzed (Participants) | 58 | 58
degrees | 13.9 (19.97) | 17.3 (20.72)

9. Secondary Outcome: Jobe Test at Visit 5 (Day 15) With Measurement of Pain
Description: This test looked for pain and weakness and was to be examined as active movement. Patients have to stand with shoulders in 90 degrees of abduction, 30 degrees of forward flexion and then internally rotating arm completely i.e., thumb pointing down. This was done to see if the patient was able to resist the clinician's attempts to depress the upper arm to look for muscle weakness.
Time Frame: Baseline vs. Day 22
Measure: Number; unit: participants
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj | Saline Inj.
Number analyzed (Participants) | 58 | 58 | 27
participants | 29 | 27 | 10

10. Secondary Outcome: Jobe Test at Visit 5 (Day 22) With Measurement of Weakness
Description: as for outcome 9
Time Frame: Baseline vs. day 22
Measure: Number; unit: participants
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj | Saline Inj.
Number analyzed (Participants) | 58 | 58 | 27
participants | 19 | 19 | 6

11. Secondary Outcome: Painful Arc Test at Visit 5 (Day 22)
Description: The amount of pain that disappeared by further abduction in the range between 60° and 120° was to be measured, with measurement of pain being positive/negative. The idea behind the test is the subacromial space in abduction becomes smaller, whereby compression of the rotator cuff and the subacromial bursa occurs (impingement test).
Time Frame: Baseline vs. day 22
Measure: Number; unit: participants
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj | Saline Inj.
Number analyzed (Participants) | 58 | 58 | 27
participants | 29 | 30 | 12

12. Secondary Outcome: Change From Baseline in DASH at Visit 5 (Day 22)
Description: The score from the questions answered on the DASH (Disaability of the Arm, Shoulder and Hand) questionnaire were evaluated on both shoulders at screening and on the target shoulder at the later visits. Any changes between the score from baseline was used to evaluate efficacy.
  The score consists of a basic questionnaire of 30 questions regarding the daily activities with the answer options from "no difficulty" (value 1) to "unable" (value 5).
  The calculation is: ((sum of values of responses/number of responses)-1) X 25. Best possible result is 0, worst possible result is 100. The score may not be calculated if there are more than 3 missing answers.
Time Frame: Baseline vs. Day 22
Measure: Mean (Standard Deviation); unit: DASH score
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj | Saline Inj.
Number analyzed (Participants) | 58 | 58 | 27
DASH score | -11.00 (13.648) | -18.03 (19.230) | -12.59 (17.698)

13. Secondary Outcome: Change From Baseline in DASH at Visit 7 (Day 105)
Description: The score from the questions answered on the DASH (Disaability of the Arm, Shoulder and Hand) questionnaire were evaluated on both shoulders at screening and on the The score consists of a basic questionnaire of 30 questions regarding the daily activities with the answer options from "no difficulty" (value 1) to "unable" (value 5).
  The calculation is: ((sum of values of responses/number of responses)-1) X 25. Best possible result is 0, worst possible result is 100. The score may not be calculated if there are more than 3 missing answers.target shoulder at the later visits. Any changes between the score from baseline was used to evaluate efficacy
Time Frame: Baseline vs. Day 105
Measure: Mean (Standard Deviation); unit: DASH score
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj | Saline Inj.
Number analyzed (Participants) | 58 | 58 | 27
DASH score | -20.91 (19.747) | -22.07 (27.697) | -19.77 (20.802)

ADVERSE EVENTS:
Time Frame: Adverse Events have been collected for 15 months between 16.Apr.2013 (first Patient in) and 23.Jun.2014 (last Patient out).
Arm/Group | Traumeel S Inj. | Fortecortin/Dexamethasone 8 mg Inj | Saline Inj.
Serious Adverse Events (participants affected / at risk) | 0/72 | 1/67 | 0/36
Other Adverse Events (participants affected / at risk) | 8/72 | 6/67 | 7/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traumeel S Inj. (N=72) | Fortecortin/Dexamethasone 8 mg Inj (N=67) | Saline Inj. (N=36)
Auricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — The event was severe and led to discontinuation of study drug after the first injection. The patient had a medical history of a previous event of auricular fibrillation since 2002. Both investigator and Heel considered the SAE as "unrelated".
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Traumeel S Inj. (N=72) | Fortecortin/Dexamethasone 8 mg Inj (N=67) | Saline Inj. (N=36)
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less